CLINICAL TRIAL: NCT00817362
Title: A Phase 2 Multicenter Study Evaluating the Efficacy and Safety of IPI-504 in Combination With Trastuzumab in Patients With Pretreated, Locally Advanced or Metastatic Human Epidermal Growth Factor Receptor 2 (HER2) Positive Breast Cancer
Brief Title: Efficacy and Safety of IPI-504 With Trastuzumab Pretreated, Locally Advanced or Metastatic HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited efficacy response observed during interim analysis.
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-07
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; HER2 Positive Breast Cancer; Metastatic Breast Cancer; Cancer of the Breast
Keywords: Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; HER2 Positive Breast Cancer; Cancer of the breast; Trastuzumab; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — tanespimycin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-504 and Trastuzumab (Experimental): IPI-504 IV infusion 300 mg/m2 once weekly in combination with trastuzumab infusion every 3 weeks. (Continuous schedule)
  Three week cycle with IPI-504 twice per week for 2 weeks and trastuzumab once per cycle followed by one week without treatment.
  Trastuzumab IV infusion 8 mg/kg as the first dose of trastuzumab, followed by trastuzumab 6 mg/kg every 3 weeks. Subjects whose last dose of trastuzumab was <4 weeks prior to study entry will receive 6 mg/kg as the first dose of trastuzumab. For all additional cycles in Stage 1, trastuzumab will be administered with the first dose of IPI-504.
  IPI-504 and trastuzumab will be administered for all cycles. Until progression or unacceptable toxicity develops.
  Interventions: Drug: IPI-504; Drug: Trastuzumab

INTERVENTIONS:
Drug: IPI-504 — IPI-504 IV infusion 300 mg/m2
Drug: Trastuzumab — Trastuzumab IV infusion 8 mg/kg as the first dose of trastuzumab, followed by trastuzumab 6 mg/kg every 3 weeks. Subjects whose last dose of trastuzumab was <4 weeks prior to study entry will receive 6 mg/kg as the first dose of trastuzumab. For all additional cycles in Stage 1, trastuzumab will be administered with the first dose of IPI-504.
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to see if IPI-504 in combination with trastuzamab is an effective treatment in HER2 positive metastatic breast cancer

DETAILED DESCRIPTION:
Recent clinical data has demonstrated that even in heavily pretreated patients with trastuzumab-refractory HER-2 positive breast cancer, targeting HER2 is efficacious.

IPI-504 is an HSP90 inhibitor and is chemically related to 17-AAG and it has been studied in a clinical trial in combination with trastuzamab and a response rate of 26% (7/27) was demonstrated in patients with pretreated, HER2-positive breast cancer. These data provide a strong scientific rationale for clinical testing of IPI-504 plus trastuzumab in patients with pretreated, locally advanced or metastatic HER2-positive breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced/metastatic breast cancer.
* HER2-expressing primary or metastatic tumor
* Two prior regimens with HER2. Trastuzumab must have been given. No limit to prior therapies
* Measurable disease with RECIST 1.1
* Clinical progression
* LVEF WNL
* ECOG 0 or 1
* Last dose of chemotherapy, radiotherapy, surgery, ablative therapy, tyrosine kinase inhibitor, ≥2 weeks
* Administration of biological therapy ≥4 weeks
* Last dose of trastuzumab must be ≥1, or ≥3 weeks prior to start, if previously administered on an every 3 week schedule.
* Resolution of toxic effects to baseline or Grade 1, except alopecia (NCI CTCAE Version 3.0
* Organ and marrow function:

  * Hemoglobin ≥8.0 g/dL
  * ANC ≥1200/µL
  * Platelets ≥75,000 /µL
  * ALT and AST ≤ 1.5 x ULN
  * Alkaline phosphatase ≤2.5 x ULN, or ≤3.0 x ULN if secondary to liver metastases.
  * Serum bilirubin WNL
  * Serum albumin ≥3.0 g/dL
  * PT, PTT ≤1.5 x ULN
  * Serum creatinine ≤1.5 x ULN
* Negative pregnancy test

Exclusion Criteria:

* Prior treatment with Hsp90 inhibitor.
* Grade 4 AE secondary to trastuzumab. Grade 3/4 infusion reactions or Grade 3/4 symptomatic heart failure
* Medication/food that is a CYP3A inhibitor or inducer.
* Hx 6 months: cardiac disease - acute coronary syndrome or unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, cirrhotic liver disease, cerebrovascular accident or significant co-morbid condition
* Grade 3 or 4 hemorrhagic event within 6 months.
* HIV positivity
* Baseline QT corrected, QTcF >470 ms
* Sinus bradycardia <50 bpm Secondary to pharmacologic therapy may enroll if stopping therapy normalizes heart rate.
* Malignancies within 3 years other than non-melanomatous skin cancers, non-muscle-invasive bladder cancer and carcinoma in situ of cervix.
* Active keratitis or keratoconjunctivitis
* Active brain metastasis (e.g., requiring therapy with steroids or radiation therapy; or with intracranial progression 4 weeks after the completion of radiation therapy) uncontrolled seizure disorder, ongoing spinal cord compression, or carcinomatous meningitis. If clinically stable brain metastasis (previously treated or untreated)are present pt is eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate overall response rate, safety, and tolerability of IPI-504 plus trastuzumab in patients with pretreated, locally advanced or metastatic HER2 positive breast cancer | After initial 20 patients are enrolled and treated for one cycle - if less that 33% of the subjects experience a dose limiting toxicity an additional 26 subjects will be enrolled

SECONDARY OUTCOMES:
Evaluate the progression-free survival (PFS) time to progression (TTP) and overall survival(OS) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Santabarbara, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (11):
- United States (10):
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Boca Raton Comphrensive Cancer Care, Boca Raton, Florida
  - Florida Cancer Research Institute, Davie, Florida
  - Peachtree Hematology-Oncology Consultants, P.C., Atlanta, Georgia
  - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Breast Center, New York, New York
  - West Cancer Clinic, Memphis, Tennessee
  - US Oncology, Dallas, Texas
- Vall d'Hebron Institute of Oncology (V.H.I.O.), Barcelona, Spain